CLINICAL TRIAL: NCT02832700
Title: Casein Glycomacropeptide in Healthy Subjects - Anti-inflammatory and Microbiome Modulating Effects
Brief Title: Casein Glycomacropeptide in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Arla Foods (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CGMPH2016
Record Dates: First submitted 2016-06-30; First posted 2016-07-14 (Estimated); Last update posted 2019-06-10 (Actual); Status verified 2016-06

CONDITIONS: Gastrointestinal Disease
Keywords: glycopeptides; dietary proteins; whey protein; caseinomacropeptide; antiinflammatories; human microbiome
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Casein glycomacropeptide (CGMP) (Active Comparator): During 4 weeks a daily oral intake of CGMP-protein-shake.
  Interventions: Dietary Supplement: Casein glycomacropeptide
- Placebo (Placebo Comparator): During 4 weeks a daily oral intake of placebo-shake consisting of milk powder.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Casein glycomacropeptide
  Arms: Casein glycomacropeptide (CGMP)
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
Casein glycomacropeptide (CGMP) has anti-inflammatory properties in experimental rodent colitis and using human in vitro inflammation models. Its use as a food ingredient has proven safe and with no influence on dietary intake. In a pilot study the investigators found, that orally administered CGMP seems to have a beneficial effect comparable to that of mesalazine in active distal ulcerative colitis.

The investigators now wish to evaluate the effects in healthy subjects by studying the anti-inflammatory and microbiome modulating properties and by assessing possible changes in gastrointestinal symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Caucasians
* Body Mass Index 18.5-25.0

Exclusion Criteria:

* Within 3 months: Acute intestinal disease (diarrhea more than 3 days in a week or bloody stools), hospital admission or antibiotic treatment.
* Chronic inflammatory disease or intestinal disease, including Crohn's disease, ulcerative colitis, celiac disease, rheumatoid arthritis or any other autoimmune joint disease, multiple sclerosis or any intestinal surgery apart from appendectomy.
* Pregnant or nursing.
* Unable to speak and understand Danish.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-06; Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with changes in systemic inflammation markers and cellular immune response | 4 weeks
  C-reactive protein, leukocyte count

SECONDARY OUTCOMES:
Number of participants with changes in the intestinal microbiome | 4 weeks
  alfa- and beta-diversity
Number of participants with changes in gastrointestinal symptoms | 4 weeks
  questionnaire

OTHER OUTCOMES:
Compliance | 4 weeks
  Number of participants with an average daily intake of above 75% of the intervention-product
Intestinal butyrate production | 4 weeks
  Number of participants with increase in daily butyrate-production

CONTACTS AND LOCATIONS:
Overall Officials: Hendrik A Vilstrup, Professor, Study Chair — University of Aarhus
Locations (1):
- Department of medicine V (Hepatology and Gastroenterology), Aarhus C, Denmark